CLINICAL TRIAL: NCT05459480
Title: The Effects of the Jigsaw Technique in Web-based Distance Education of Nursing Students: a Randomized Controlled Trial
Brief Title: The Jigsaw Technique in Nursing Education
Acronym: jigsaw
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ayşe Aydınlı, RN,PhD, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SuleymanDUn
Record Dates: First submitted 2022-07-05; First posted 2022-07-15 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-07

CONDITIONS: Nursing Student; Education
Keywords: Nursing student; Motivation; Jigsaw method; Self-Confidence; distance education; Academic Achievement

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Students will be given information about the study, but not in which group they are included. Thus, blinding will be ensured.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Online training was continued according to the jigsaw technique for a total of 6 weeks, two hours a week. In the first week, 6 subgroups of 6 people were created.
  Sub-topics of the physical examination course were shared according to the systems to these groups, called the main group.
  In the first week, it was aimed for the groups to get to know each other and the first lesson was used for that. In the second week, the students in the main group researched the sub-topics of the unit given to them and formed a new group by coming together with students who were researching the same subject. This group was called the expert group. In the third and fourth weeks, expert groups continued their studies to reinforce the subject.
  In the fifth and sixth group the students returned to their main groups and explained the subjects they had learned in the expert groups to their main group. Students were expected to teach each other all parts of the unit in their main groups.
  Interventions: Other: the jigsaw technique in web-based distance education
- Control Group (No Intervention): The subjects were explained by the instructor with the traditional e-teaching method and as in the intervention group, the lectures were conducted online for two hours a week for 6 weeks. At the end of each week, the relevant course documents were shared with the students. At the end of the sixth week, the post-tests of the learning motivation and self-confidence scales were applied in the control group simultaneously with the intervention group. In addition, an academic achievement test was applied.

INTERVENTIONS:
Other: the jigsaw technique in web-based distance education — The online training for the intervention group continued for a total of 6 weeks according to the jigsaw technique.
  Arms: Intervention Group

SUMMARY:
Aim: This study aimed to determine the effect of the jigsaw technique on students' self-confidence, learning motivation, and academic success in physical examination e-teaching according to systems as a randomized controlled trial. The volunteering students were divided into two groups, intervention and control groups, according to a randomization made with a computer program. The Jigsaw Technique was applied to the intervention group, while the control group received the traditional learning method. To avoid interaction between the groups, the lessons in the intervention and control groups were conducted by different instructors. Prior to the application, data collection tools were applied to the intervention and control groups as a pre-test.

DETAILED DESCRIPTION:
Aim: This study aimed to determine the effect of the jigsaw technique on students' self-confidence, learning motivation, and academic success in physical examination e-teaching according to systems as a randomized controlled trial. The volunteering students were divided into two groups, intervention and control groups, according to a randomization made with a computer program. The Jigsaw Technique was applied to the intervention group, while the control group received the traditional learning method. To avoid interaction between the groups, the lessons in the intervention and control groups were conducted by different instructors.

Intervention Group; Starting from the week following the pre-test application, online training was continued according to the jigsaw technique for a total of 6 weeks, two hours a week, for the intervention group. In the first week, 6 subgroups of 6 people were created. Sub-topics of the physical examination course were shared according to the systems to these groups, called the main group, and the course documents were shared with the students.

In the first week, it was aimed for the groups to get to know each other and the first lesson was used for that. A responsible student was determined for each main group, names were given to the groups. In the second week, the students in the main group researched the sub-topics of the unit given to them and formed a new group by coming together with students who were researching the same subject. This group was called the expert group. In these groups, the students shared their course information and studied the subject by exchanging ideas to explain the subject they were working on to their friends. In the third and fourth weeks, expert groups continued their studies to reinforce the subject.

In the fifth and sixth groups, the students returned to their main groups and explained the subjects they had learned in the expert groups to their main group. Students were expected to teach each other all parts of the unit in their main groups. In the intervention group, the instructor only fulfilled the role of a guide and explained subjects that the students had difficulties understanding. At the end of the six weeks, the learning motivation and self-confidence scales were re-administered as a post-test. In addition, an academic achievement test was applied.

Control Group; The subjects were explained by the instructor with the traditional e-teaching method and as in the intervention group, the lectures were conducted online for two hours a week for 6 weeks. At the end of each week, the relevant course documents were shared with the students. At the end of the sixth week, the post-tests of the learning motivation and self-confidence scales were applied in the control group simultaneously with the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Having volunteered to participate in the study
* Being a first-year nursing student
* Taking the course diagnostics of health

Exclusion Criteria:

* Not having volunteered to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Learning Motivation Scale | 6 weeks
  The scale was developed by Noe and Wilk in 1993. It is a 5-point Likert scale (1: I totally disagree, 2: I disagree, 3: I neither agree nor disagree, 4: I agree, and 5: I totally agree) and consists of 17 items. The total scale score ranges from 17 to 85. It is expected that as the mean score increases the motivation to learn takes a positive direction. The Cronbach Alpha reliability coefficient of the scale was determined as 0.90.
Self-Confidence Scale | 6 weeks
  It was developed by Akın (2007) to determine the existing self-confidence levels of individuals and consists of 33 items. It is a 5-point Likert scale and is scores as 1: Never, 2: Sometimes, 3: Often, 4: Generally, and 5: Always. The scale consists of two subdimensions; internal self-confidence and external self-confidence. The Cronbach Alpha reliability coefficient of the scale was determined as 0.83.
Academic Achievement Test; | 6 weeks
  The academic achievement test used in the study was prepared by an expert lecturer. The tests consists of 25 multiple-choice questions. The test duration is determined as 30 minutes. With this test, it is aimed to determine the knowledge level of the students for the Diagnostics of Health course.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Çetinkaya Uslusoy, Study Chair — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned to publish the research data in the form of an article.

REFERENCES:
- [Background] Sanaie N, Vasli P, Sedighi L, Sadeghi B. Comparing the effect of lecture and Jigsaw teaching strategies on the nursing students' self-regulated learning and academic motivation: A quasi-experimental study. Nurse Educ Today. 2019 Aug;79:35-40. doi: 10.1016/j.nedt.2019.05.022. Epub 2019 May 11. PMID 31102795
- [Background] Leyva-Moral JM, Riu Camps M. Teaching research methods in nursing using Aronson's Jigsaw Technique. A cross-sectional survey of student satisfaction. Nurse Educ Today. 2016 May;40:78-83. doi: 10.1016/j.nedt.2016.02.017. Epub 2016 Feb 24. PMID 27125153
- [Background] Eycan O, Ulupinar S. Nurse instructors' perception towards distance education during the pandemic. Nurse Educ Today. 2021 Dec;107:105102. doi: 10.1016/j.nedt.2021.105102. Epub 2021 Aug 18. PMID 34482209
- [Background] Singh HK, Joshi A, Malepati RN, Najeeb S, Balakrishna P, Pannerselvam NK, Singh YK, Ganne P. A survey of E-learning methods in nursing and medical education during COVID-19 pandemic in India. Nurse Educ Today. 2021 Apr;99:104796. doi: 10.1016/j.nedt.2021.104796. Epub 2021 Feb 6. PMID 33607513